CLINICAL TRIAL: NCT03152227
Title: Evaluation of Integrated Agriculture and Nutrition Sensitive Interventions for the African Chicken Genetic Gains (ACGG) Program in Ethiopia
Brief Title: Nutrition-sensitive Agricultural Interventions for Ethiopia
Acronym: ATONU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: The International Livestock Research Institute (ILRI) (Other); Addis Continental Institute of Public Health (Other); Food, Agriculture and Natural Resources Policy Analysis Network (Unknown)
Responsible Party: Principal Investigator, Wafaie Fawzi, Dr., Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSPH-16-0912
Record Dates: First submitted 2016-11-11; First posted 2017-05-12 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Dietary Modification; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACGG & ATONU (Experimental): ACGG high-producing chicks to households along with provision of technical input on production and ATONU Nutrition sensitive BCC on poultry-specific aspects of nutrition, WASH, women's empowerment, and use of income combined with home gardening.
  Interventions: Other: ACGG; Behavioral: BCC
- ACGG only (Active Comparator): ACGG high-producing chicks to households along with provision of technical input on production
  Interventions: Other: ACGG
- Control (No Intervention): ACGG eligible households in non-ACGG villages receiving standard of care agricultural and health services as provided in Ethiopia

INTERVENTIONS:
Other: ACGG — 50 high-producing chicks to households along with provision of technical input on production
  Other Names: Chicken intensification
  Arms: ACGG & ATONU; ACGG only
Behavioral: BCC — Nutrition sensitive BCC on poultry-specific aspects of nutrition, WASH, women's empowerment, and use of income combined with home gardening.
  Other Names: ATONU
  Arms: ACGG & ATONU

SUMMARY:
This study aims at evaluating the impact of integrating nutrition sensitive behavioral change communication (BCC) in the context of increased household production of chicken and eggs on women and children diet.

DETAILED DESCRIPTION:
The Agriculture to Nutrition (ATONU) Project, led by the Food, Agriculture and Natural Resources Policy Analysis Network (FANRPAN), aims to develop, implement, and evaluate nutrition-sensitive interventions within the context of existing agricultural programs with the goal of improving the nutritional status of women of reproductive age and young children, particularly in the first 1000 days of life. Specifically, ATONU will implement a nutrition sensitive intervention in collaboration with the ACGG Program. ACGG is evaluating the agricultural productivity of high-producing chicken genotypes in Ethiopia and will be providing 20-30 chickens to small-scale chicken-producing households for an 18-month on-farm evaluation. These households will also be provided with regular technical input on good chicken production practices, and ACGG investigators will aim to reach women as well as men in participating households.

ATONU will implement an additional nutrition-sensitive intervention among ACGG households that will use behavior change communication (BCC) to encourage consumption of chicken products (meat and eggs); good water, sanitation, and hygiene (WASH) practices in poultry production; use of income from sale of chicken products to improve nutrition; empowerment of women in decision-making around chicken production and sale; and home gardening of nutrient-dense vegetables to improve dietary quality within the household. Qualitative work is supporting development of this intervention.

ACGG's intervention to increase chicken production may improve the nutritional status of women and children through increasing access to chicken meat and eggs for household consumption and empowering women by giving them access to income, which could be used for purchase of other nutrient-dense foods. However, increasing production and income alone may not necessarily translate into improved diets or nutritional outcomes. ATONU's intervention will specifically encourage the use of chicken products and income to provide nutritious diets for women of reproductive age, emancipated minors and young children through extensive nutrition behavior change communication. Further, recognizing that lack of availability of nutrient-dense foods in local markets may be an important barrier to a diverse and nutritious diet, the home gardening component of ATONU's intervention seeks to increase the availability of nutrient-dense vegetables at household level.

The ACGG program is operating in diverse agroecologies in Ethiopia. Within its target areas, the program listed villages in which chicken production was an important activity and, from this list, randomly selected villages in which to implement its intervention. In a subset of these ACGG villages, ATONU will implement its intervention. As a result, there will be two groups of ACGG villages: those receiving only the poultry production intervention, and those receiving the poultry production intervention coupled with ATONU's nutrition-sensitive intervention. Allocation of ACGG villages to one of these two groups will be done randomly. Investigators will evaluate the nutritional impact of these two interventions among smallholder chicken-producing households in Ethiopia. Specifically, investigators will use the two groups of villages described above and a third group of ACGG-eligible villages that ACGG did not choose for intervention to conduct a cluster-randomized controlled trial with the goal of evaluating the effect of the ACGG and ATONU interventions on maternal and child diets, nutritional status, and health.

ELIGIBILITY:
Inclusion Criteria:

Households in one of the two ACGG treatment arms will be eligible for inclusion if they meet all of the following criteria:

1. Are participating in the ACGG program
2. Have at least one woman of reproductive age (18-49 years at enrollment) or emancipated minor (girl aged 15 to less than 18 years)
3. Plan to remain in the study area throughout the study duration
4. Provide informed consent.

Households in the control arm will be eligible for inclusion if they meet all of the following criteria:

1. Meet the criteria for participating in the ACGG program, namely, they have produced chickens for at least two years and are currently keeping no more than 50 chickens with interest to expand production in the future
2. Have at least one woman of reproductive age (18-49 years at enrollment) or emancipated minor (girl aged 15 to less than 18 years)
3. Plan to remain in the study area throughout the study duration
4. Provide informed consent.

Exclusion Criteria:

* Households will be excluded if they fail to meet any of the criteria listed above

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2117 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Diet quality for women and emancipated minors using the standard FAO/FANTA MDD-W dietary diversity score questionnaire, | 18 months
  For each woman or emancipated minor in each study group (ACGG alone, ACGG plus ATONU, and Control), the number of food groups consumed in the previous day, out of the 10 food groups listed on the standard FAO/FHI360 MDD-W dietary diversity score questionnaire

SECONDARY OUTCOMES:
Diet quality for young children using the standard dietary diversity score questionnaire developed by the by Food and Nutrition Technical Assistance Project and Academy for Educational Development. | 18 months
  For each young child in each study group (ACGG alone, ACGG plus ATONU, and Control), the number of food groups consumed in the previous day, out of the 8 groups listed (FGI-8) on the standard dietary diversity score questionnaire developed by Food and Nutrition Technical Assistance Project and Academy for Educational Development. The dietary diversity score is based on consumption of 8 food groups in the past 24 hours.
Anemia in women and emancipated minors as defined by hemoglobin (Hb) levels cut off points of Hb < 12 g/dl for non pregnant women and Hb < 11g/dl for pregnant women | 18 months
  Defining Anemia in women and emancipated minors in the three study groups (ACGG alone, ACGG plus ATONU, and Control) using Hb cut off adjusted for altitude as per the WHO 2011 guidelines
Anemia in children as defined by hemoglobin (Hb) levels cut off points of Hb < 11 g/dl | 18 months
  Defining Anemia in children in the three study groups (ACGG alone, ACGG plus ATONU, and Control) using Hb cut off adjusted for altitude as per the WHO 2011 guidelines
Body Mass Index (BMI in kg/m^2 ) for women and emancipated minors in the three study groups (ACGG alone, ACGG plus ATONU, and Control) | 18 months
  For each woman and emancipated minor, BMI will be calculated by dividing body weight(kg) by the square of participant height (m^2). BMI values will be analyzed as continuous data.
Growth in height for children (Height for Age) in the three study groups (ACGG alone, ACGG plus ATONU, and Control) | 18 months
  Height for age will be assessed and presented as Z scores as per the WHO children height for age growth charts for boys and girls
Weight in children (Weight for Age) in the three study groups (ACGG alone, ACGG plus ATONU, and Control) | 18 months
  Weight for age in children will be assessed and presented as Z scores as per the WHO children weight for age charts for boys and girls

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, DrPH,MBBS, Principal Investigator — Harvard School of Public Health (HSPH); Yemane Berhane, PhD, Principal Investigator — Addis Continental Institute of Public Health
Locations (1):
- Addis Continental Institute of Public Health (ACIPH), Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
data sharing agreement in progress

REFERENCES:
- [Background] Balarajan Y, Ramakrishnan U, Ozaltin E, Shankar AH, Subramanian SV. Anaemia in low-income and middle-income countries. Lancet. 2011 Dec 17;378(9809):2123-35. doi: 10.1016/S0140-6736(10)62304-5. Epub 2011 Aug 1. PMID 21813172
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Iannotti LL, Lutter CK, Bunn DA, Stewart CP. Eggs: the uncracked potential for improving maternal and young child nutrition among the world's poor. Nutr Rev. 2014 Jun;72(6):355-68. doi: 10.1111/nure.12107. Epub 2014 May 7. PMID 24807641
- [Background] Lee AC, Katz J, Blencowe H, Cousens S, Kozuki N, Vogel JP, Adair L, Baqui AH, Bhutta ZA, Caulfield LE, Christian P, Clarke SE, Ezzati M, Fawzi W, Gonzalez R, Huybregts L, Kariuki S, Kolsteren P, Lusingu J, Marchant T, Merialdi M, Mongkolchati A, Mullany LC, Ndirangu J, Newell ML, Nien JK, Osrin D, Roberfroid D, Rosen HE, Sania A, Silveira MF, Tielsch J, Vaidya A, Willey BA, Lawn JE, Black RE; CHERG SGA-Preterm Birth Working Group. National and regional estimates of term and preterm babies born small for gestational age in 138 low-income and middle-income countries in 2010. Lancet Glob Health. 2013 Jul;1(1):e26-36. doi: 10.1016/S2214-109X(13)70006-8. Epub 2013 Jun 25. PMID 25103583
- [Background] Leroy JL, Frongillo EA. Can interventions to promote animal production ameliorate undernutrition? J Nutr. 2007 Oct;137(10):2311-6. doi: 10.1093/jn/137.10.2311. PMID 17885016
- [Background] Marquis GS, Habicht JP, Lanata CF, Black RE, Rasmussen KM. Breast milk or animal-product foods improve linear growth of Peruvian toddlers consuming marginal diets. Am J Clin Nutr. 1997 Nov;66(5):1102-9. doi: 10.1093/ajcn/66.5.1102. PMID 9356526
- [Background] Olofin I, McDonald CM, Ezzati M, Flaxman S, Black RE, Fawzi WW, Caulfield LE, Danaei G; Nutrition Impact Model Study (anthropometry cohort pooling). Associations of suboptimal growth with all-cause and cause-specific mortality in children under five years: a pooled analysis of ten prospective studies. PLoS One. 2013 May 29;8(5):e64636. doi: 10.1371/journal.pone.0064636. Print 2013. PMID 23734210
- [Background] Ruel MT, Alderman H; Maternal and Child Nutrition Study Group. Nutrition-sensitive interventions and programmes: how can they help to accelerate progress in improving maternal and child nutrition? Lancet. 2013 Aug 10;382(9891):536-51. doi: 10.1016/S0140-6736(13)60843-0. Epub 2013 Jun 6. PMID 23746780
- [Background] Stevens GA, Finucane MM, Paciorek CJ, Flaxman SR, White RA, Donner AJ, Ezzati M; Nutrition Impact Model Study Group (Child Growth). Trends in mild, moderate, and severe stunting and underweight, and progress towards MDG 1 in 141 developing countries: a systematic analysis of population representative data. Lancet. 2012 Sep 1;380(9844):824-34. doi: 10.1016/S0140-6736(12)60647-3. Epub 2012 Jul 5. PMID 22770478
- [Background] Sudfeld CR, McCoy DC, Danaei G, Fink G, Ezzati M, Andrews KG, Fawzi WW. Linear growth and child development in low- and middle-income countries: a meta-analysis. Pediatrics. 2015 May;135(5):e1266-75. doi: 10.1542/peds.2014-3111. Epub 2015 Apr 6. PMID 25847806
- [Background] Victora CG, Adair L, Fall C, Hallal PC, Martorell R, Richter L, Sachdev HS; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: consequences for adult health and human capital. Lancet. 2008 Jan 26;371(9609):340-57. doi: 10.1016/S0140-6736(07)61692-4. PMID 18206223
- [Derived] Passarelli S, Ambikapathi R, Gunaratna NS, Madzorera I, Canavan CR, Noor RA, Tewahido D, Berhane Y, Sibanda S, Sibanda LM, Madzivhandila T, Munthali BLM, McConnell M, Sudfeld C, Davison K, Fawzi W. The role of chicken management practices in children's exposure to environmental contamination: a mixed-methods analysis. BMC Public Health. 2021 Jun 8;21(1):1097. doi: 10.1186/s12889-021-11025-y. PMID 34103022
- [Derived] Ambikapathi R, Passarelli S, Madzorera I, Canavan CR, Noor RA, Abdelmenan S, Tewahido D, Tadesse AW, Sibanda L, Sibanda S, Munthali B, Madzivhandila T, Berhane Y, Fawzi W, Gunaratna NS. Men's nutrition knowledge is important for women's and children's nutrition in Ethiopia. Matern Child Nutr. 2021 Jan;17(1):e13062. doi: 10.1111/mcn.13062. Epub 2020 Aug 4. PMID 32755057
- [Derived] Passarelli S, Ambikapathi R, Gunaratna NS, Madzorera I, Canavan CR, Noor AR, Worku A, Berhane Y, Abdelmenan S, Sibanda S, Munthali B, Madzivhandila T, Sibanda LM, Geremew K, Dessie T, Abegaz S, Assefa G, Sudfeld C, McConnell M, Davison K, Fawzi W. A Chicken Production Intervention and Additional Nutrition Behavior Change Component Increased Child Growth in Ethiopia: A Cluster-Randomized Trial. J Nutr. 2020 Oct 12;150(10):2806-2817. doi: 10.1093/jn/nxaa181. PMID 32652012